CLINICAL TRIAL: NCT02515630
Title: A Phase 2, Open-label, Translational Biology Study of Momelotinib in Transfusion-Dependent Subjects With Primary Myelofibrosis (PMF) or Post-polycythemia Vera or Post-essential Thrombocythemia Myelofibrosis (Post-PV/ET MF)
Brief Title: Momelotinib in Transfusion-Dependent Adults With Primary Myelofibrosis (PMF) or Post-polycythemia Vera or Post-essential Thrombocythemia Myelofibrosis (Post-PV/ET MF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-352-1672
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Primary Myelofibrosis (PMF); Post-polycythemia Vera (Post-PV) Myelofibrosis; Postessential Thrombocythemia (Post-ET) Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Momelotinib (Experimental): MMB for 24 weeks (± 7 days)
  Interventions: Drug: MMB

INTERVENTIONS:
Drug: MMB — Momelotinib (MMB) tablet administered orally once daily
  Other Names: GS-0387; CYT387

SUMMARY:
This study will evaluate the transfusion independence response rate in transfusion-dependent adults with myelofibrosis after treatment with momelotinib (MMB).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of PMF or Post PV/ET-MF
* Requires myelofibrosis therapy, in the opinion of the investigator
* High risk OR intermediate-2 risk defined by dynamic international prognostic scoring system (DIPSS) OR intermediate-1 risk defined by DIPSS and associated with symptomatic splenomegaly and/or hepatomegaly
* Transfusion dependent at baseline, defined as ≥ 4 U red blood cell (RBC) transfusion in the 8 weeks prior to first dose of MMB
* Acceptable organ function as evidenced by the following:

  * Platelet Count ≥ 50 x 10^9/L
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3 x upper limit of normal (ULN) or AST or ALT ≤ 5 x ULN if liver is involved by disease process as judged by the investigator
  * Serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance of ≥ 60 mL/min
  * Direct bilirubin ≤ 2.0 x ULN
* Life expectancy of > 24 weeks
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Lactating females must agree to discontinue nursing before MMB administration
* Able to understand and willing to sign the informed consent form

Key Exclusion Criteria:

* Prior splenectomy
* Splenic irradiation within 3 months prior to the first dose of MMB
* Prior treatment with MMB
* Known positive status of human immunodeficiency virus (HIV)
* Chronic active or acute viral hepatitis A, B, or C infection (testing required for hepatitis B and C), or hepatitis B or C carrier
* Use of strong cytochrome P450 3A4 (CYP3A4) inducer within 2 weeks prior to the first dose of MMB
* Uncontrolled intercurrent illness per protocol
* Treatment with a Janus kinase (JAK) inhibitor within 21 days of the planned first dose of MMB
* Presence of peripheral neuropathy ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Unwilling or unable to undergo a MRI per requirements in the study protocol
* Unwilling to consent to genomics sampling

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- United States (12):
  - Phoenix, Arizona
  - Los Angeles, California
  - Orange, California
  - Jacksonville, Florida
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Houston, Texas
- Toronto, Ontario, Canada

REFERENCES:
- [Derived] Harrison CN, Mesa R, Talpaz M, Gupta V, Gerds AT, Perkins A, Goh YT, Fox ML, McLornan D, Palmer J, Foltz L, Vannucchi A, Koschmieder S, Passamonti F, Lee SE, Ellis C, Strouse B, Gonzalez Carreras FJ, Oh ST. Longitudinal Assessment of Transfusion Intensity in Patients With JAK Inhibitor-Naive or -Experienced Myelofibrosis Treated With Momelotinib. Clin Lymphoma Myeloma Leuk. 2025 Mar;25(3):199-211. doi: 10.1016/j.clml.2024.10.001. Epub 2024 Oct 16. PMID 39516087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled transfusion-dependent myelofibrosis patients at oncology centers in the United States and Canada. Following completion of the 24-week study period, patients who were benefiting had the option to continue maintenance momelotinib treatment in an open-label extension study (NCT02124746).
Groups:
- Momelotinib (MMB): Subjects received oral MMB at a starting dose of 200 mg once daily for 24 weeks (± 7 days) on study.
Period: Overall Study
Arm/Group | Momelotinib (MMB)
Started | 41
Completed | 25
Not Completed | 16
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 4
Not completed — Physician Decision | 4
Not completed — Death | 2
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Transfusion Independence Responders: Subjects who became transfusion independent by Week 24
- Transfusion Independence Non-Responders: Subjects who did not become transfusion independent by Week 24
- Total: Total of all reporting groups
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.0) | 72 (7.5) | 70 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 8 | 18 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 2 | 3
  White | 11 | 25 | 36
  Not Permitted | 1 | 0 | 1
  Other | 1 | 0 | 1
Spleen Volume [Mean (Standard Deviation); unit: cm^3] | 2132.2 (1439.5) | 2018.1 (1248.5) | 2057.1 (1299.8)
Total Symptom Score [Mean (Standard Deviation); unit: units on a scale] — Total symptom score was assessed using the modified MPN-SAF TSS Version 2, an 8-item questionnaire developed to assess symptom burden and quality of life in patients with MPN. The modified MPN-SAF TSS contained 8 questions, 7 of which were summed to generate the score (the included questions related to tiredness, early satiety, abdominal discomfort, night sweats, itching, bone pain, and pain under the ribs on the left side). Each question is scored on a scale of 0-10, where higher numbers indicate more severe symptoms. For this study, the TSS scale ranges from 0 to 70.
  units on a scale | 19.00 (16.14) | 21.73 (13.97) | 20.73 (14.65)
RBC Units Transfused within 8 weeks prior to Enrollment [Mean (Standard Deviation); unit: Units of red blood cell] | 5 (1.9) | 7 (2.2) | 6 (2.3)
Hepcidin [Median (Inter-Quartile Range); unit: nM] | 22.0 [9.6 to 33.9] | 42.4 [27.4 to 64.9] | 36.6 [18.6 to 48.5]
Serum iron [Median (Inter-Quartile Range); unit: ug/dL] | 96.0 [56.0 to 123.0] | 127.0 [105.0 to 174.0] | 119.0 [84.0 to 165.0]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 8.5 [7.6 to 9.4] | 7.8 [7.3 to 8.4] | 8.0 [7.4 to 8.8]
Total iron binding capacity [Median (Inter-Quartile Range); unit: ug/dL] | 214.5 [178.0 to 239.0] | 201.0 [181.0 to 269.0] | 205.0 [181.0 to 253.0]
Reticulocytes [Median (Inter-Quartile Range); unit: cells*10^6/uL] | 0.096 [0.055 to 0.127] | 0.067 [0.039 to 0.094] | 0.071 [0.043 to 0.102]
Reticulocytes/erythrocytes [Median (Inter-Quartile Range); unit: %] | 3.5 [1.8 to 4.3] | 2.2 [1.4 to 3.2] | 2.4 [1.7 to 3.5]
Erythropoietin [Median (Inter-Quartile Range); unit: mIU/mL] | 238.7 [63.3 to 499.4] | 88.1 [27.5 to 287.6] | 109.8 [30.0 to 493.0]
Erythrocytes [Median (Inter-Quartile Range); unit: cells*10^6/uL] | 3.0 [2.8 to 3.2] | 2.8 [2.6 to 3.3] | 2.9 [2.6 to 3.2]
Hematocrit [Median (Inter-Quartile Range); unit: %] | 27.5 [25.0 to 28.0] | 24.0 [22.0 to 28.0] | 25.0 [22.0 to 28.0]
Ferritin [Median (Inter-Quartile Range); unit: ng/mL] | 605.9 [372.7 to 1018.5] | 1259.4 [441.6 to 2321.5] | 1008.9 [441.6 to 1634.5]
Soluble transferrin receptor [Median (Inter-Quartile Range); unit: mg/L] | 2.5 [1.6 to 5.8] | 1.3 [0.7 to 2.1] | 1.6 [1.0 to 2.5]
Transferrin saturation [Median (Inter-Quartile Range); unit: %] | 43.0 [33.0 to 54.0] | 56.5 [47.5 to 63.0] | 53.0 [42.0 to 60.0]
Unsaturated iron binding capacity [Median (Inter-Quartile Range); unit: ug/dL] | 113.5 [30.0 to 151.0] | 81.0 [37.0 to 124.0] | 92.0 [37.0 to 127.0]
Platelets [Median (Inter-Quartile Range); unit: cells*10^3/uL] | 190.5 [72.0 to 262.0] | 134.0 [106.0 to 211.0] | 146.0 [106.0 to 222.0]
Leukocytes [Median (Inter-Quartile Range); unit: cells*10^3/uL] | 6.4 [3.8 to 7.7] | 8.5 [4.5 to 11.4] | 6.4 [4.5 to 11.0]
Blasts [Median (Inter-Quartile Range); unit: %] | 0 [NA to NA] — No blasts measured | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0]
Liver Iron Content [Median (Inter-Quartile Range); unit: mg/g] | 2.4 [1.6 to 4.0] | 4.2 [2.6 to 11.3] | 3.5 [2.3 to 6.4]
%pSTAT Stimulated CD3+/4+ T cell [Median (Inter-Quartile Range); unit: %] | 85.1 [76.9 to 87.1] | 77.8 [60.3 to 91.5] | 79.8 [67.6 to 88.2]
%pSTAT %tSTAT Stimulated CD3+/4+ T cell Ratio [Median (Inter-Quartile Range); unit: ratio] | 0.9 [0.9 to 1.0] | 0.8 [0.6 to 1.0] | 0.9 [0.7 to 1.0]
C-Reactive Protein [Median (Inter-Quartile Range); unit: mg/dL] | 0.7 [0.4 to 1.8] | 1.8 [0.6 to 4.5] | 1.2 [0.6 to 3.8]

OUTCOME MEASURES:

1. Primary Outcome: Transfusion Independence Response by Week 24
Description: The percentage of subjects who became transfusion independent for ≥ 12 weeks at any time on study. A subject was considered transfusion independent on study if no RBC transfusion occurred in any 12-week period during the 24-week treatment period.
Time Frame: From baseline to Week 24
Population: Assessed in the Safety Analysis Set, which includes all subjects who received ≥ 1 dose of momelotinib. Note that 6 subjects discontinued prior to Week 12 and could not be evaluated over the minimum period required for assessment of the endpoint (12 weeks).
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Groups:
- Total: All enrolled subjects
Arm/Group | Total
Number analyzed (Participants) | 41
percentage of subjects | 34.1 [22.0 to 48.1]

2. Secondary Outcome: Transfusion Response Rate by Week 24
Description: The percentage of subjects who became transfusion independent for ≥ 8 weeks, defined as no RBC transfusions for at least an 8-week period at any time on study.
Time Frame: From baseline to Week 24
Population: Assessed in the Safety Analysis Set, which includes all subjects who received ≥ 1 dose of momelotinib. Note that 3 subjects discontinued prior to Week 8 and could not be evaluated over the minimum period required for assessment of the endpoint (8 weeks).
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Total
Number analyzed (Participants) | 41
percentage of subjects | 39.0 [26.2 to 53.1]

3. Secondary Outcome: Splenic Response Rate at Week 24
Description: The percentage of subjects who achieved a ≥ 35% reduction in spleen volume from baseline as measured by MRI at Week 24.
Time Frame: Measured at Week 24
Population: Assessed in the Safety Analysis Set, which includes all subjects who received ≥ 1 dose of momelotinib. Note that spleen volume at Week 24 was not available for 15 subjects.
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Total
Number analyzed (Participants) | 41
percentage of subjects | 12.2 [4.9 to 23.9]

4. Secondary Outcome: Response Rate in Total Symptom Score (TSS) at Week 24
Description: The percentage of subjects achieving a ≥ 50% reduction from baseline in TSS at Week 24, as measured by the modified Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPNSAF TSS) diary. Total symptom score was assessed using the modified MPN-SAF TSS Version 2, an 8-item questionnaire developed to assess symptom burden and quality of life in patients with MPN. The modified MPN-SAF TSS contained 8 questions, 7 of which were summed to generate the score (the included questions related to tiredness, early satiety, abdominal discomfort, night sweats, itching, bone pain, and pain under the ribs on the left side). Each question is scored on a scale of 0-10, where higher numbers indicate more severe symptoms. For this study, the TSS scale ranges from 0 to 70. The questionnaire was completed daily on an electronic diary device.
Time Frame: Measured at Week 24
Population: There were 3 subjects with missing TSS at baseline who were excluded from the analysis. Note that of the 38 subjects evaluated, 17 were missing Week 24 TSS assessments.
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Total
Number analyzed (Participants) | 38
percentage of subjects | 15.8 [7.1 to 28.8]

5. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Change From Baseline in Hepcidin Daily Change
Description: Hepcidin daily change (in nM) was calculated as the predose value subtracted from the 6 hours postdose value at each study visit. Daily hepcidin change at the baseline visit was the difference between 2 values obtained 6 hours apart. No momelotinib was administered on that day.
Time Frame: At baseline, Day 1, Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: nM
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
nM
  Baseline | -1.7 [-2.1 to 4.7] | 0.1 [-3.3 to 4.5] | 0.0 [-3.3 to 4.6]
  Day 1 | -4.8 [-10.2 to -1.4] | -11.2 [-16.0 to -5.8] | -8.6 [-14.4 to -3.3]
  Week 2 | -4.9 [-9.1 to -0.4] | -6.7 [-11.3 to -1.2] | -6.3 [-9.2 to -0.7]
  Week 4 | -2.6 [-8.5 to 0.1] | -7.4 [-9.6 to -0.9] | -5.4 [-9.6 to 0.1]
  Week 8 | -2.9 [-7.3 to -0.9] | -5.2 [-17.7 to 2.1] | -4.4 [-10.9 to -0.6]
  Week 12 | -1.4 [-6.8 to 0.7] | -5.7 [-8.7 to -0.9] | -4.1 [-8.4 to 0.5]
  Week 16 | -0.4 [-6.4 to 0.7] | -4.3 [-15.1 to 1.9] | -2.7 [-8.5 to 1.1]
  Week 20 | 0.0 [-6.6 to 4.2] | -7.8 [-12.5 to -1.9] | -5.3 [-9.0 to 1.5]
  Week 24 | -1.0 [-4.6 to 0.1] | -1.8 [-7.8 to 0.1] | -1.4 [-6.0 to 0.1]

6. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Trough Hepcidin
Description: Median hepcidin at trough was assessed predose at each study visit.
Time Frame: At baseline, Day 1, Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: nM
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
nM
  Baseline | 22.0 [9.6 to 33.9] | 42.4 [27.4 to 64.9] | 36.6 [18.6 to 48.5]
  Day 1 | 19.7 [5.5 to 30.8] | 43.7 [29.9 to 58.7] | 36.5 [22.4 to 48.0]
  Week 2 | 25.1 [14.6 to 29.7] | 52.1 [37.4 to 61.2] | 38.4 [25.8 to 57.6]
  Week 4 | 19.8 [13.7 to 30.8] | 46.4 [39.1 to 57.1] | 37.6 [19.8 to 51.9]
  Week 8 | 16.6 [10.1 to 29.2] | 51.7 [39.9 to 59.4] | 35.5 [16.9 to 52.7]
  Week 12 | 21.3 [10.9 to 30.4] | 44.7 [23.3 to 53.9] | 30.4 [15.6 to 44.8]
  Week 16 | 16.9 [7.1 to 29.0] | 51.9 [43.7 to 62.9] | 34.5 [17.1 to 51.9]
  Week 20 | 13.4 [4.5 to 27.4] | 44.2 [31.5 to 49.7] | 27.5 [13.4 to 44.3]
  Week 24 | 15.5 [4.9 to 28.8] | 51.5 [27.9 to 60.2] | 28.4 [14.2 to 45.2]

7. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Serum Iron
Description: Percent change from baseline in serum iron, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 4.5 [-14.6 to 73.2] | 5.9 [-10.3 to 31.0] | 5.9 [-11.8 to 39.6]
  Week 4 | 39.8 [1.8 to 108.1] | 5.7 [-16.2 to 33.3] | 13.3 [-12.7 to 57.8]
  Week 8 | 9.3 [-23.6 to 44.0] | 5.4 [-15.6 to 42.0] | 6.4 [-18.2 to 44.0]
  Week 12 | 3.0 [-25.2 to 73.2] | 14.3 [3.1 to 35.1] | 12.8 [-7.9 to 39.4]
  Week 16 | -15.5 [-20.3 to 56.6] | 16.5 [-19.3 to 30.7] | 8.9 [-19.4 to 30.7]
  Week 20 | -11.1 [-17.8 to 41.7] | 9.9 [-7.4 to 28.1] | 1.9 [-17.8 to 34.6]
  Week 24 | -8.1 [-20.4 to 45.1] | -5.1 [-24.3 to 31.1] | -6.6 [-22.9 to 37.4]

8. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Hemoglobin
Description: Percent change from baseline in hemoglobin, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change in from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change in from baseline
  Week 2 | 12.8 [0.0 to 20.3] | 9.2 [0.0 to 26.3] | 9.9 [0.0 to 20.4]
  Week 4 | 8.3 [1.4 to 15.9] | 6.3 [-1.2 to 20.6] | 6.9 [-1.2 to 20.6]
  Week 8 | 12.4 [4.8 to 27.7] | 0.4 [-7.7 to 14.2] | 5.6 [-6.3 to 19.1]
  Week 12 | 15.6 [5.3 to 25.3] | 4.5 [-12.5 to 13.4] | 7.5 [-4.8 to 17.4]
  Week 16 | 12.3 [4.8 to 32.9] | 0.6 [-9.5 to 15.0] | 10.2 [-6.3 to 19.7]
  Week 20 | 13.1 [5.3 to 28.9] | 6.9 [-7.1 to 17.3] | 7.4 [-3.9 to 17.9]
  Week 24 | 10.0 [-2.1 to 29.4] | 5.8 [-1.3 to 14.4] | 7.9 [-1.4 to 17.6]

9. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Total Iron Binding Capacity
Description: Percent change from baseline in total iron binding capacity, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 4.5 [0.4 to 13.6] | 2.0 [-5.5 to 8.9] | 2.8 [-1.6 to 10.1]
  Week 4 | 6.7 [-2.5 to 15.7] | 1.5 [-9.6 to 10.7] | 2.2 [-5.6 to 11.0]
  Week 8 | 4.9 [-2.7 to 10.3] | 0.6 [-7.4 to 13.7] | 2.4 [-6.6 to 11.5]
  Week 12 | 6.6 [-3.9 to 12.6] | 2.4 [-5.9 to 20.2] | 6.6 [-5.5 to 15.1]
  Week 16 | 4.5 [-3.2 to 9.8] | 1.5 [-10.0 to 14.2] | 3.6 [-5.3 to 11.3]
  Week 20 | 15.5 [3.4 to 22.1] | 5.5 [-11.6 to 15.4] | 10.6 [1.6 to 17.2]
  Week 24 | 7.3 [3.6 to 15.8] | 0.5 [-8.4 to 10.7] | 5.5 [-5.9 to 13.0]

10. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Reticulocytes
Description: Percent change from baseline in reticulocytes, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 33.6 [-6.7 to 67.5] | -9.6 [-26.0 to 26.4] | 2.9 [-23.6 to 36.2]
  Week 4 | 11.8 [4.0 to 40.7] | 5.5 [-32.7 to 46.4] | 7.5 [-29.3 to 43.5]
  Week 8 | 30.0 [13.2 to 35.0] | -16.0 [-30.6 to 28.4] | 15.6 [-24.5 to 31.0]
  Week 12 | 15.8 [-6.3 to 45.1] | -9.5 [-34.5 to 33.3] | 4.8 [-17.3 to 44.2]
  Week 16 | 31.2 [-22.1 to 58.5] | 8.8 [-24.0 to 35.5] | 18.3 [-23.1 to 45.6]
  Week 20 | 34.0 [-35.6 to 70.4] | 7.7 [-48.6 to 27.7] | 16.3 [-44.8 to 48.1]
  Week 24 | 29.9 [11.5 to 58.3] | -0.6 [-32.0 to 67.8] | 24.1 [-12.0 to 58.4]

11. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Reticulocytes/Erythrocytes%
Description: Percent change from baseline in reticulocytes/erythrocytes%, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 30.0 [-16.7 to 42.6] | -16.3 [-30.1 to 23.6] | -8.0 [-28.1 to 36.4]
  Week 4 | 8.2 [-7.0 to 20.4] | 1.5 [-36.3 to 29.6] | 4.1 [-29.9 to 26.5]
  Week 8 | 12.4 [-5.6 to 33.3] | -11.1 [-35.3 to 27.8] | 0.0 [-21.2 to 27.8]
  Week 12 | 3.6 [-11.1 to 16.7] | 0.0 [-31.6 to 42.3] | 0.0 [-29.4 to 42.3]
  Week 16 | 4.4 [-22.9 to 33.3] | 18.7 [-30.0 to 50.0] | 7.8 [-29.0 to 41.7]
  Week 20 | 2.2 [-34.3 to 21.4] | 14.6 [-43.8 to 46.2] | 11.1 [-42.1 to 46.2]
  Week 24 | 2.2 [-2.9 to 24.1] | -7.8 [-34.2 to 72.6] | -2.6 [-11.8 to 72.2]

12. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Erythropoietin
Description: Percent change in erythropoietin at Weeks 8 and 20. The baseline erythropoietin value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 8 and 20
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 8 | -30.8 [-55.6 to -6.8] | -8.1 [-47.7 to 31.3] | -24.5 [-55.4 to 29.4]
  Week 20 | -45.0 [-63.4 to -2.0] | 8.5 [-16.2 to 82.9] | -4.4 [-60.2 to 32.5]

13. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Erythrocytes
Description: Percent change from baseline in erythrocytes, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 5.2 [0.0 to 20.0] | 3.4 [-6.1 to 12.1] | 3.4 [-6.1 to 16.7]
  Week 4 | 6.7 [-8.8 to 13.3] | 3.6 [-3.6 to 21.5] | 3.8 [-3.7 to 16.0]
  Week 8 | 3.6 [-2.0 to 23.3] | 0.0 [-13.1 to 13.0] | 3.0 [-6.1 to 22.9]
  Week 12 | 3.1 [-3.6 to 26.7] | 3.6 [-13.8 to 11.4] | 3.4 [-10.0 to 23.1]
  Week 16 | 0.0 [-8.8 to 26.7] | -6.9 [-9.2 to 6.5] | -2.9 [-8.8 to 12.0]
  Week 20 | -3.3 [-12.0 to 26.7] | -3.4 [-13.8 to 7.7] | -3.4 [-12.1 to 12.2]
  Week 24 | -8.0 [-9.7 to 26.7] | 3.3 [-7.1 to 11.4] | 0.0 [-9.7 to 19.2]

14. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Hematocrit
Description: Percent change from baseline in hematocrit, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 8.9 [-4.3 to 18.5] | 4.0 [-4.8 to 11.1] | 4.5 [-4.8 to 16.1]
  Week 4 | 7.4 [-5.6 to 10.7] | 0.0 [-4.3 to 21.4] | 3.4 [-4.3 to 20.0]
  Week 8 | 11.1 [3.6 to 25.9] | -1.7 [-14.6 to 14.8] | 4.0 [-7.1 to 17.9]
  Week 12 | 7.1 [-3.1 to 30.8] | 1.8 [-13.0 to 14.8] | 3.6 [-8.0 to 18.2]
  Week 16 | 5.9 [-3.2 to 28.6] | -4.2 [-8.3 to 8.2] | 3.8 [-7.7 to 10.7]
  Week 20 | 7.1 [-3.2 to 26.9] | 0.0 [-12.0 to 4.3] | 0.0 [-7.9 to 12.8]
  Week 24 | 8.0 [-3.6 to 28.6] | 2.3 [-9.1 to 9.1] | 4.5 [-8.3 to 14.8]

15. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Ferritin
Description: Percent change from baseline in ferritin, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 11.6 [-11.2 to 35.9] | 8.8 [-0.2 to 25.3] | 8.8 [-7.4 to 31.0]
  Week 4 | 19.1 [-6.8 to 32.9] | 8.3 [-3.5 to 38.8] | 13.6 [-3.8 to 35.3]
  Week 8 | 4.0 [-24.1 to 15.9] | 30.4 [-5.6 to 38.7] | 16.7 [-10.1 to 32.5]
  Week 12 | -0.6 [-11.2 to 11.3] | 26.4 [4.3 to 52.0] | 11.3 [-10.0 to 31.0]
  Week 16 | 0.1 [-24.6 to 8.0] | 21.6 [0.7 to 100.9] | 6.7 [-8.7 to 30.9]
  Week 20 | 3.5 [-42.9 to 23.1] | 13.6 [-10.0 to 74.6] | 7.0 [-33.6 to 61.8]
  Week 24 | -14.2 [-40.2 to 6.6] | 15.4 [-20.7 to 59.7] | 1.4 [-27.2 to 42.6]

16. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Soluble Transferrin Receptor
Description: Percent change from baseline in soluble transferrin receptor, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 4.0 [-14.7 to 18.1] | -4.9 [-12.8 to 6.3] | -4.8 [-14.1 to 16.7]
  Week 4 | -1.4 [-7.0 to 26.2] | 8.8 [-16.6 to 31.5] | 0.7 [-16.6 to 30.9]
  Week 8 | 6.7 [-15.3 to 24.0] | 11.0 [-15.1 to 37.2] | 7.4 [-15.3 to 28.4]
  Week 12 | 0.8 [-18.3 to 13.5] | 11.1 [2.0 to 38.8] | 10.7 [-13.5 to 23.9]
  Week 16 | -0.1 [-17.3 to 19.2] | 14.9 [-9.1 to 32.3] | 1.3 [-9.1 to 27.3]
  Week 20 | -1.8 [-11.2 to 10.6] | -0.7 [-7.4 to 21.2] | -1.2 [-11.2 to 14.1]
  Week 24 | -3.5 [-15.5 to 10.0] | 19.7 [-24.2 to 30.8] | -1.8 [-16.7 to 26.1]

17. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Transferrin Saturation
Description: Percent change from baseline in transferrin saturation, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 2.4 [-15.2 to 52.1] | 13.5 [-6.7 to 35.6] | 10.3 [-8.3 to 44.1]
  Week 4 | 36.4 [4.2 to 75.0] | 9.7 [-17.2 to 36.7] | 10.5 [-4.8 to 45.8]
  Week 8 | 9.5 [-21.7 to 33.3] | -5.0 [-23.1 to 26.2] | -3.1 [-22.4 to 29.7]
  Week 12 | 11.9 [-18.6 to 52.9] | 16.4 [-3.8 to 26.3] | 14.1 [-18.3 to 26.7]
  Week 16 | -7.2 [-22.2 to 40.7] | -13.5 [-24.6 to 33.3] | -10.4 [-24.6 to 40.7]
  Week 20 | -2.5 [-20.7 to 36.4] | -20.8 [-40.4 to 8.3] | -13.3 [-31.9 to 9.3]
  Week 24 | -8.3 [-22.1 to 23.7] | -20.8 [-31.7 to 25.0] | -11.9 [-25.0 to 25.0]

18. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Unsaturated Iron Binding Capacity
Description: Percent change from baseline in unsaturated iron binding capacity, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 0.0 [-39.4 to 13.2] | -5.1 [-31.1 to 14.6] | 0.0 [-31.5 to 13.2]
  Week 4 | -4.0 [-24.3 to 1.9] | 0.0 [-35.7 to 34.0] | -1.0 [-25.3 to 28.1]
  Week 8 | 6.4 [-25.0 to 28.0] | 0.0 [-40.2 to 31.8] | 0.0 [-29.9 to 28.4]
  Week 12 | 2.9 [-17.4 to 31.4] | -18.4 [-33.6 to 7.0] | -1.6 [-32.3 to 21.4]
  Week 16 | 4.3 [-22.4 to 34.7] | 0.0 [-49.2 to 21.4] | 2.6 [-35.6 to 30.5]
  Week 20 | 16.5 [-12.0 to 62.8] | 5.1 [-39.8 to 44.0] | 14.2 [-15.9 to 46.7]
  Week 24 | 12.0 [2.5 to 32.2] | 6.9 [-35.7 to 64.9] | 12.0 [-11.3 to 64.9]

19. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Platelets
Description: Percent change from baseline in platelets, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 21.4 [-25.4 to 48.9] | -24.4 [-41.8 to 6.3] | -9.5 [-37.4 to 32.1]
  Week 4 | 0.0 [-25.5 to 49.1] | -29.7 [-43.7 to -4.1] | -26.3 [-35.9 to 9.6]
  Week 8 | 19.7 [-1.3 to 57.2] | -33.6 [-48.2 to 3.3] | -12.0 [-40.3 to 23.0]
  Week 12 | 24.1 [7.9 to 83.7] | -27.7 [-49.0 to -11.5] | -11.4 [-39.9 to 27.3]
  Week 16 | 17.8 [2.3 to 80.0] | -26.1 [-48.0 to -6.2] | -6.2 [-31.3 to 30.8]
  Week 20 | 31.0 [-6.9 to 41.4] | -36.2 [-67.1 to -10.7] | -14.3 [-37.8 to 34.3]
  Week 24 | 38.9 [-15.4 to 78.3] | -22.5 [-52.1 to -8.8] | -15.3 [-30.2 to 60.9]

20. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Leukocytes
Description: Percent change from baseline in leukocytes, where the baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 4, 8, 12, 16, 20 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 11.6 [-10.0 to 42.9] | -24.9 [-34.8 to 1.5] | -14.9 [-29.8 to 11.4]
  Week 4 | 6.8 [-18.3 to 38.6] | -4.7 [-26.4 to 11.4] | 0.7 [-21.1 to 19.8]
  Week 8 | 34.3 [11.6 to 57.1] | -0.9 [-18.9 to 13.4] | 8.9 [-14.0 to 30.5]
  Week 12 | 8.0 [5.4 to 48.4] | -15.4 [-35.5 to 22.9] | 5.4 [-24.2 to 38.7]
  Week 16 | 42.0 [14.6 to 53.7] | -6.7 [-26.9 to 27.0] | 15.2 [-14.3 to 45.7]
  Week 20 | 44.7 [13.0 to 70.5] | -27.5 [-42.1 to 24.8] | 16.3 [-32.8 to 49.1]
  Week 24 | 53.0 [0.2 to 75.3] | 18.3 [-35.4 to 42.9] | 27.1 [-26.4 to 63.4]

21. Secondary Outcome: Change in Markers of Iron Metabolism and Anemia - Blasts
Description: Change from baseline in % blasts at Weeks 2 and 4. The baseline % blasts value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2 and 4
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | 0 [NA to NA] — No blasts measured | 3.0 [3.0 to 3.0] | 3.0 [3.0 to 3.0]
  Week 4 | 0 [NA to NA] — No blasts measured | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

22. Secondary Outcome: Change in Liver Iron Content
Description: Percent change from baseline in liver iron content assessed by MRI. The baseline value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: Measured at Week 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline | 4.7 [-18.4 to 25.0] | 53.3 [20.6 to 86.2] | 22.3 [-6.0 to 71.7]

23. Secondary Outcome: Change in Pharmacodynamics Biomarker - pSTAT3
Description: Percent change in %pSTAT stimulated CD3+/4+ T cell at Day 1 (postdose), Week 4 and Week 24. The baseline value is defined as the last predose value from the baseline period prior to or on the date of first dose of momelotinib administration (Day 1 predose).
Time Frame: On Day 1 and at Weeks 4 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Day 1 - 2 hours postdose | -15.8 [-34.2 to -11.6] | -13.5 [-24.4 to -7.6] | -14.3 [-27.7 to -9.6]
  Day 1 - 4 hours postdose | -17.1 [-23.4 to -8.1] | -10.6 [-30.6 to -2.4] | -12.8 [-27.3 to -6.6]
  Day 1 - 6 hours postdose | -9.0 [-16.9 to -4.0] | -4.3 [-16.9 to 0.3] | -7.1 [-16.9 to -2.2]
  Week 4 - predose | -0.9 [-2.0 to 1.8] | -2.9 [-5.5 to 17.7] | -2.0 [-5.5 to 17.7]
  Week 4 - 2 hours postdose | -18.9 [-21.9 to -6.6] | -20.0 [-25.7 to -7.4] | -20.0 [-25.7 to -6.6]
  Week 4 - 4 hours postdose | -19.8 [-30.4 to -8.8] | -14.1 [-28.7 to -6.1] | -14.1 [-30.4 to -6.1]
  Week 4 - 6 hours postdose | -12.1 [-29.0 to -1.5] | -9.1 [-12.9 to 4.9] | -9.1 [-19.0 to 4.9]
  Week 24 - predose | -4.6 [-22.9 to 0.1] | -0.3 [-7.9 to 5.1] | -2.8 [-22.9 to 5.1]
  Week 24 - 2 hours postdose | -31.2 [-51.2 to -18.0] | -10.7 [-28.4 to -10.1] | -22.7 [-48.2 to -10.7]
  Week 24 - 4 hours postdose | -30.6 [-65.8 to -17.6] | -14.4 [-22.6 to -12.9] | -22.6 [-50.1 to -14.1]
  Week 24 - 6 hours postdose | -17.0 [-33.2 to -13.4] | -10.1 [-10.2 to -4.9] | -13.4 [-24.8 to -10.1]

24. Secondary Outcome: Change in Pharmacodynamics Biomarker - pSTAT3/tSTAT3 Ratio
Description: Percent change in %pSTAT/%tSTAT Stimulated CD3+/4+ T cell ratio at Day 1 (postdose), Week 4 and Week 24. The baseline value is defined as the last predose value from the baseline period prior to or on the date of first dose of momelotinib administration (Day 1 predose).
Time Frame: On Day 1 and at Weeks 4 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Day 1 - 2 hours postdose | -13.2 [-38.9 to -11.5] | -15.5 [-23.2 to 2.5] | -13.4 [-26.3 to -3.2]
  Day 1 - 4 hours postdose | -9.6 [-23.2 to -0.5] | -9.7 [-28.0 to -2.3] | -9.7 [-23.9 to -2.3]
  Day 1 - 6 hours postdose | -9.1 [-17.2 to -5.7] | -3.7 [-12.1 to 3.7] | -4.6 [-13.7 to 1.7]
  Week 4 - predose | 0.5 [-5.2 to 31.8] | 5.0 [-4.3 to 39.8] | 4.8 [-5.2 to 39.8]
  Week 4 - 2 hours postdose | -14.3 [-17.5 to 20.3] | -9.1 [-22.6 to 9.6] | -13.2 [-22.6 to 20.3]
  Week 4 - 4 hours postdose | 3.0 [-32.9 to 118.3] | -13.4 [-23.7 to 23.9] | -13.4 [-31.5 to 38.1]
  Week 4 - 6 hours postdose | 12.5 [-29.4 to 56.0] | -6.1 [-17.1 to 32.8] | -6.1 [-20.5 to 56.0]
  Week 24 - predose | -5.7 [-17.4 to -3.7] | -3.5 [-8.8 to -2.8] | -4.4 [-17.4 to -2.8]
  Week 24 - 2 hours postdose | -18.7 [-22.3 to -15.4] | -7.6 [-22.1 to -2.6] | -16.2 [-22.3 to -2.6]
  Week 24 - 4 hours postdose | -21.4 [-27.1 to -14.3] | -11.5 [-15.4 to -9.6] | -15.4 [-27.0 to -11.5]
  Week 24 - 6 hours postdose | -18.4 [-22.8 to -11.1] | -6.5 [-9.0 to -5.1] | -11.1 [-20.0 to -5.1]

25. Secondary Outcome: Change in Inflammatory Markers - C-Reactive Protein (CRP)
Description: Percent change in C-reactive protein at Weeks 2, 12 and 24. The baseline C-reactive protein value is defined as the last value from the baseline period prior to or on the date of first dose of momelotinib administration (Baseline visit).
Time Frame: At Weeks 2, 12 and 24
Measure: Median (Inter-Quartile Range); unit: % Change from baseline
Arm/Group | Transfusion Independence Responders | Transfusion Independence Non-Responders | Total
Number analyzed (Participants) | 14 | 27 | 41
% Change from baseline
  Week 2 | -68.7 [-75.6 to -43.5] | -53.7 [-76.8 to -18.5] | -55.6 [-76.3 to -29.5]
  Week 12 | -67.8 [-73.1 to -28.2] | -43.4 [-59.6 to 22.6] | -48.9 [-70.1 to -15.6]
  Week 24 | -59.8 [-79.1 to -44.8] | -47.1 [-68.4 to 65.3] | -54.8 [-73.8 to -30.7]

ADVERSE EVENTS:
Time Frame: From the first dose of momelotinib until 30 days following the last dose.
Description: All adverse events summarized were treatment-emergent, defined as any adverse event with an onset date on or after the momelotinib start date and no later than 30 days after permanent discontinuation of momelotinib or any adverse event leading to premature discontinuation of momelotinib.
Arm/Group | Momelotinib (MMB)
All-Cause Mortality (participants affected / at risk) | 3/41
Serious Adverse Events (participants affected / at risk) | 14/41
Other Adverse Events (participants affected / at risk) | 36/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Momelotinib (MMB) (N=41)
Anemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Presyncope (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 1
Pyrexia (General disorders) | 1
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Momelotinib (MMB) (N=41)
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 5
Fatigue (General disorders) | 8
Chills (General disorders) | 3
Urinary tract infection (Infections and infestations) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 7
Night sweats (Skin and subcutaneous tissue disorders) | 3
Blood creatinine increased (Investigations) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Contusion (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 4
Pollakiuria (Renal and urinary disorders) | 3
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Pharmacokinetics parameters were removed as an analysis endpoint in the SAP due to the sparse PK samples collection.

Change in circulating cytokine and inflammatory markers were limited to CRP as an analysis endpoint in the SAP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Most restrictive: Site may not present or publish results of Trial without advance written notice of Sponsor or two years after completion of Trial at all participating sites. Site must submit all proposed publications or presentations to Sponsor for review. Sponsor can review communications prior to public release and embargo trial results communications for a period between 75 and 180 days from submission to Sponsor for review. Sponsor has right to request Site remove Confidential Information.

DOCUMENTS (2):
  • Study Protocol (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT02515630/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT02515630/SAP_001.pdf